CLINICAL TRIAL: NCT04323605
Title: Implementation of an Assistance Program for Outpatients Following an Allogeneic Hematopoietic Stem-cell Transplant: Pilot Feasibility Study
Brief Title: Assistance Program for Outpatients Following an Allogeneic Hematopoietic Stem-cell Transplant
Acronym: AMA-ALLO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: RC31/16/8771
Record Dates: First submitted 2020-03-24; First posted 2020-03-26 (Actual); Last update posted 2020-12-03 (Actual); Status verified 2020-12

CONDITIONS: Hematologic Neoplasms
Keywords: allogeneic hematopoietic stem-cell transplant; outpatient assistance; "navigation" nurse
MeSH Terms: conditions — Hematologic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- outpatient assistance program (Experimental)
  Interventions: Other: Outpatient assistance program for transplant patients (AMA-ALLO) based on a "navigation" nurse

INTERVENTIONS:
Other: Outpatient assistance program for transplant patients (AMA-ALLO) based on a "navigation" nurse — Integration of a post-transplant "navigation" nurse starting at the first post-transplant consultation (starting from D100 +/- 10 days post-transplant). Different times for post-transplant telephone monitoring (every week for the first 2 months, then every 15 days for the next 3 months then once a month for 7 months)

SUMMARY:
After the initial monitoring period during hospitalization and isolation, patients with recent transplants are regularly monitored in monthly consultations but are still fragile, immunosuppressed and undergoing many treatments. The implementation of an outpatient assistance program for transplant patients should be feasible and allow for the improvement in medical-psycho-social care for the patients during this fragile and risky period, improve the satisfaction and quality of life for these transplant patients and assist in their socio-professional and familial reintegration.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients over 18 years of age
* Having received an allogeneic hematopoietic stem-cell transplant
* In full remission
* Outpatients
* Having given their informed consent for the participation in the outpatient assistance program with a navigation nurse (AMA-ALLO) at the first post-transplant consultation (starting on Day 100 +/- 10 days post-transplant i.e., when the patient passes the initial post-transplant monitoring period in hospitalization (conventional or by day) to the monitoring period in monthly medical consultations) and continuing for 12 months
* Affiliated with the social security system

Exclusion Criteria:

* Transplant patients not having given their informed consent for inclusion in AMA-ALLO
* Hospitalized or non-outpatient transplant patients
* Post-transplant patients in cytological relapse
* Patients under a legal regime of adult protection (guardianship, curatorship, etc.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-01 (Estimated); Primary Completion 2022-01 (Estimated); Study Completion 2022-02 (Estimated)

PRIMARY OUTCOMES:
Rate of patients with all the navigation nurse intervention files received at 100% | 12 months
  Rate of patients with all the navigation nurse intervention files received at 100%.
  A file is received at 100% if the 4 following tasks are fully completed:
  1. - patient called by nurse (and response from the patient at the set telephone appointment)
  2. - completion of medical-psycho-social questionnaire (AMA-ALLO phone call form) by nurse with the patient's responses
  3. - information and transmission of questionnaire results by nurse to the transplant physician
  4. - physician/nurse decision for potential intervention (specialized consultation, consultation with the transplant physician, hospitalization, modification of treatments, additional exams to carry out, etc.)

SECONDARY OUTCOMES:
Rate of refusal for participation in the study | 12 months
  Rate of patients who refused participating in the study
Rate of ineligibility of the navigation nurse intervention files | 12 months
  Rate of ineligibility of the navigation nurse intervention files (a single incomplete task out of 4 per intervention file renders the file ineligible)
Quality of life for transplant patients | Baseline
  Quality of life for transplant patients is assessed with the Functional Assessment of Cancer Therapy--Leukemia (FACT-Leu) questionnaire version 4. Fo each question, the 5 modality answers are: 0=not all, 1= a little bit, 2=somewhat, 3=quite a bit, 4=very much
Quality of life for transplant patients | 6 months
  Quality of life for transplant patients is assessed with the Functional Assessment of Cancer Therapy--Leukemia (FACT-Leu) questionnaire version 4. Fo each question, the 5 modality answers are: 0=not all, 1= a little bit, 2=somewhat, 3=quite a bit, 4=very much
Quality of life for transplant patients | 12 months
  Quality of life for transplant patients is assessed with the Functional Assessment of Cancer Therapy--Leukemia (FACT-Leu) questionnaire version 4. Fo each question, the 5 modality answers are: 0=not all, 1= a little bit, 2=somewhat, 3=quite a bit, 4=very much

CONTACTS AND LOCATIONS:
Overall Officials: Anne HUYNH, MD, Principal Investigator — University hospital of Toulouse
Locations (1):
- Toulouse University Hospital, Toulouse, France